CLINICAL TRIAL: NCT03941613
Title: Stereotactic-EEG Guided Radio-frequency Thermocoagulation Versus Anterior Temporal Lobectomy for Mesial Temporal Lobe Epilepsy With Hippocampus Sclerosis
Brief Title: SEEG Guided RF-TC v.s. ATL for mTLE With HS
Acronym: STARTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018011021001
Record Dates: First submitted 2019-04-23; First posted 2019-05-08 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Epilepsy, Temporal Lobe
Keywords: temporal lobe epilepsy; hippocampus sclerosis (HS); radiofrequency thermocoagulation (RF-TC); cognitive status
MeSH Terms: conditions — Epilepsy, Temporal Lobe | interventions — Anterior Temporal Lobectomy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anterior temporal lobectomy (Experimental): surgical treatment for mTLE
  Interventions: Procedure: Anterior temporal lobectomy
- SEEG guided RF-TC (Active Comparator): SEEG recording and minimal invasive treatment for mTLE
  Interventions: Procedure: SEEG guided RF-TC

INTERVENTIONS:
Procedure: SEEG guided RF-TC — SEEG implantation after evaluation, record the interictal and ictal EEG, and perform RF-TC after the localization confirmation.
  Arms: SEEG guided RF-TC
Procedure: Anterior temporal lobectomy — classical surgical treatment for mesial temporal lobe epilepsy, including the resection of neocortex for 5.5cm in non dominant hemisphere or 4.5cm in dominant hemisphere
  Arms: Anterior temporal lobectomy

SUMMARY:
Mesial temporal lobe epilepsy (mTLE) is the most classical subtype of temporal lobe epilepsy, which is the indication of surgical intervention after evaluation. Until now, anterior temporal lobectomy (ATL) is still the recommended treatment for mTLE. However, evidences are accumulated including post ATL tetartanopia and memory deterioration and new minimized invasive treatments are introduced. Stereotactic EEG (SEEG) guided radio-frequency thermocoagulation (RF-TC) is one of the option with lower seizure freedom but with higher neurological function reservation. This study is aiming at comparison of the efficacy and safety between SEEG guided RF-TC and classical ATL in the treatment of mTLE.

DETAILED DESCRIPTION:
Nowadays, more and more patients received SEEG implantation for the evaluation of intractable seizures. SEEG is not only a diagnostic method to locate the origin of the epileptic seizures but also a media to treat or to cure this disease. Using radiofrequency thermocoagulation, we are able to coagulate some part of the brain guided by SEEG. However, until now, we don't have high level evidence for the efficacy and safety of RF-TC. In our resent series, we found the 1 year seizure free rate of mTLE patients after RF-TC is about 80% without any notable complication.

In this trail, we will compare the efficacy as well as the safety of anterior temporal lobectomy with RF-TC for the mTLE patients, including the 1 year Engel class, perioperative complications, cognitive function, visual field, etc. Thus we can provide more high level evidence on the usage of SEEG guided RF-TC on mTLE patients.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of drug resistant epilepsy

At least one or more anti-epileptic drugs (AEDs) regular administered for more than 2 years, one of which was either Dilantin, Tegretol, Carbatrol, or Trileptal used in appropriate doses, have failed due to inefficacy, not intolerance

Persistence of disabling seizures at least 3 times per 3 months or greater, and once or more in recent 1 month

14 years or older at enrollment

Simple and complex partial seizures, with or without secondarily generalized seizures beginning in childhood or later, with or without febrile convulsions earlier

Auras that occur in isolation and are not primary sensory other than olfactory or gustatory

I.Q. of greater than 70

Hippocampal atrophy on MRI T1 imaging with increased ipsilateral mesial signal on T2 imaging

Interictal EEG shows focal or lateralized spikes on temporal, frontal zone, or sphenoid electrode

Ictal EEG onset is focal or lateralized on the ipsilateral side

Ipsilateral temporal focal hypometabolism on PET

Must be agreed by a consensus of ipsilateral mesial temporal origin by a multidisciplinary discussion

Must be able to understand and speak Mandarin

Exclusion criteria:

A history of serious cerebral insult after the age of 5

A progressive neurological disorder; mental retardation (I.Q. less than 70)

Psychogenic seizures

Focal neurological deficits other than memory disturbances

Any unexplained focal or lateralized neurological deficits other than memory dysfunction.

Temporal neocortical or extratemporal lesions on MRI

Psychosis, current or recent substance abuse, suicidality, anorexia, or psychogenic seizures

Severe systemic diseases

Unequivocal focal extratemporal EEG slowing or interictal spikes

Lesions on MRI outside of the mesial temporal area

Diffuse unilateral or bilateral hypometabolism on positron emission tomography (PET)

Contralateral or extratemporal ictal onset

Persistent extratemporal, or predominant contralateral focal interictal spikes or slowing, or generalized interictal spikes

Patient who was included in any clinical trial

Pregnancy

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 1 year
  Full scaled Wechsler Adult Intelligence Quality IV Chinese edition (WAIS-IV-C), or Wechsler Children Intelligence Quality IV Chinese edition (WCIS-IV-C) Higher values represent a better outcome.

SECONDARY OUTCOMES:
Seizure freedom | 1 year
  Engel classification at 1 year
Visual field | 1 year
  Visual field examination
Number of participants with procedure related complications | 1 year
  Postoperative stroke with or without symptoms (by MRI); Postoperative intracranial bleeding with or without symptoms (by MRI); Postoperative intracranial infection; Postoperative wound infection; Postoperative subcutaneous dropsy.
Quality of life after treatment | 1 year
  Quality of Life in Epilepsy 89 (QOLIE-89) for adults (aged from 17-60), and Quality of Life in Epilepsy 89 (QOLIE-48) for children (aged from 14-16)
Average hospitalization expenses | 1 month after surgery
  Whole expenses of each group of patients

CONTACTS AND LOCATIONS:
Overall Officials: Guoguang Zhao, Doctor, Study Director — Xuanwu hospital, CCMU
Locations (1):
- Xuanwu Hospital, Capital Medical University., Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The baseline information and follow-up data are available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 1 year after the last follow-up.
Access Criteria: PI of any of Epilepsy center

REFERENCES:
- [Derived] Shan Y, Shi J, Wang T, Chen S, Feng T, Yin L, Ren L, Wei P, Yang Y, Wang H, Zhao G. Optimized stereoelectroencephalography-guided thermocoagulation versus anterior temporal lobectomy in mesial temporal epilepsy: A pilot randomized controlled study. J Adv Res. 2025 Jun 19:S2090-1232(25)00451-5. doi: 10.1016/j.jare.2025.06.042. Online ahead of print. PMID 40543839
- [Derived] Wang YH, Chen SC, Wei PH, Yang K, Fan XT, Meng F, Du JL, Ren LK, Shan YZ, Zhao GG. Stereotactic EEG-guided radiofrequency thermocoagulation versus anterior temporal lobectomy for mesial temporal lobe epilepsy with hippocampal sclerosis: study protocol for a randomised controlled trial. Trials. 2021 Jun 29;22(1):425. doi: 10.1186/s13063-021-05378-3. PMID 34187524